CLINICAL TRIAL: NCT03257059
Title: Breakfast Consumption and Its Effects on Glycemic, Insulinemic and Non-Esterified Fatty Acids Responses
Acronym: BEGIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JeyaKumar Henry (Other Government)
Collaborators: General Mills (Industry)
Responsible Party: Sponsor-Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Organization: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2017/00537
Record Dates: First submitted 2017-08-09; First posted 2017-08-22 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Glycemic Response
MeSH Terms: interventions — Breakfast

STUDY DESIGN:
Intervention Model Description: Randomised, crossover study with two treatments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breakfast (Experimental): Subject given standardized breakfast (glutinous rice) to test blood glucose response
  Interventions: Other: Breakfast
- No breakfast (Experimental): Subject not given breakfast to test blood glucose response
  Interventions: Other: No Breakfast

INTERVENTIONS:
Other: Breakfast — Glutinous rice (75 grams of available carbohydrate)
  Arms: Breakfast
Other: No Breakfast — No food to be served in the morning
  Arms: No breakfast

SUMMARY:
The aim of this study is to determine whether eating breakfast or having no breakfast has subsequent beneficial health effects, specifically in relation to glycemic response throughout the day and postprandial insulin and non-esterified fatty acids (NEFA) responses 6 hours after breakfast/lunch.

DETAILED DESCRIPTION:
This will be a randomised, crossover study with two treatments in total. 1.) Subjects given with breakfast, 2.) Subjects not given breakfast. Each of the two test visits will last for approximately 9 hour (spanning over 3 days), during which the following will take place: On Day 1, subjects will come to have the continuous glucose monitoring (CGMS) system inserted. CGMS will be used to measure 24 hour blood glucose concentrations. On Day 2, an indwelling catheter will be inserted into the ante cubital fossa or forearm vein of one arm and will be kept patent. One fasting blood sample (baseline; 4 milliliters of venous blood) will be collected. Participants with breakfast treatment will then consume the test meal within 15 minutes. Subsequently, blood samples will be taken at 15, 30, 45, 60, 90, 120, 150 and 180 minutes.At time 180 minutes, participants will be given a standardized lunch to be consumed within 30 minutes. Blood samples will be taken after lunch at 210, 240, 270, 300, 330 and 360 minutes. On Day 3, subjects will need to come for removal of the CGMS sensor. Subjects will come to the CNRC again for the 2nd test visit, with at least 3 days wash-out in-between visits.

ELIGIBILITY:
Inclusion Criteria:

* Chinese males
* BMI above 23.0 kg/m2
* Age between 40-65 years
* Normal blood pressure (<140/90 mmHg)
* Fasting blood glucose of ≥5.6 mmol/L
* Self-reported regular breakfast consumers

Exclusion Criteria:

* Have known glucose-6-phosphate dehydrogenase (G6PD) deficiency
* major chronic disease such as heart disease, cancer or diabetes mellitus
* taking insulin or drugs known to affect glucose metabolism
* Intentionally restrict food intake
* major medical or surgical event requiring hospitalization within the preceding 3 months
* Have taken antibiotics for 3 months before the study period
* Smoking
* Overnight shift workers
* Any known food allergy (eg. anaphylaxis to peanuts)
* Having active Tuberculosis (TB) or currently receiving treatment for TB
* Any known Chronic infection or known to suffer from or have previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV)
* Being a member of the research team or their immediate family members. Immediate family member is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* Enrolled in a concurrent research study judged not to be scientifically or medically compatible with the study of the CNRC.

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Glycemic response | 1.5 days
  Using continuous glucose monitoring system
Insulin response | 6 hours
  Postprandial after treatment
Non-esterified fatty acids (NEFA) response | 6 hours
  Postprandial after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No